CLINICAL TRIAL: NCT01143467
Title: Relationship Between Mitochondrial Dysfunction and Fatique in Cancer Patients Following External Beam Radiation Therapy
Status: Completed | Type: Observational
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100128; 10-NR-0128
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2015-11-06

CONDITIONS: Cancer; Fatigue
Keywords: Fatigue; Mitochondria; Mitochondrial Abnormality; Oxidative Stress; Gene Expression; Prostate Cancer
MeSH Terms: conditions — Neoplasms; Fatigue; Prostatic Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Fatigue is a very common early and late side effect of cancer treatment, including radiation therapy. The cause of fatigue is poorly understood, making it hard to diagnose and treat. More research is necessary to understand why patients receiving cancer treatment experience fatigue. Changes in mitochondria, parts of body cells that help provide energy to the cell, may contribute to fatigue. Researchers are interested in looking at blood chemicals and mitochondrial genes of cancer patients to study those associated with fatigue.

Objectives:

- To study the relationship between fatigue and the effects of cancer treatment.

Eligibility:

* Men at least 18 years of age who have been diagnosed with localized prostate cancer and are scheduled to receive external beam radiation therapy.
* Participants on study 09-NR-0088, Molecular-Genetic Correlates of Fatigue in Cancer Patients Receiving External Beam Radiation Therapy, are also eligible.

Design:

* This study requires three outpatient visits to the NIH Clinical Center.
* Participants will be seen before they start radiation treatment, at the middle of treatment, and at the end of treatment. Each visit will take less than 30 minutes to complete.
* Participants will complete questionnaires that ask about fatigue and depression.
* Participants will provide blood samples for research testing and potential HIV testing.
* No treatment will be provided as part of this protocol.

DETAILED DESCRIPTION:
Fatigue is a common early and chronic adverse effect of radiation but its correlates and prevalence are poorly understood. Over 40% of cancer patients receive radiation therapy during the management of their disease. While external beam intensity modulated radiation therapy (EBRT/IMRT) successfully increases disease-free survival rates and life expectancy, ionizing radiation leads to increased treatment-related adverse effects including fatigue. Multidimensional causes and mechanisms of cancer-related fatigue remain unclear, and early biomarkers prognostic for radiation-induced fatigue have not been identified.

There is evidence that an increase in reactive oxygen species (ROS) formation will cause cellular damage resulting in dysfunction to mitochondria. ROS are considered one of the major direct causes of ionizing radiation-induced damage, resulting in a number of adverse effects (e.g. fatigue, nausea, vomiting, diarrhea, peripheral neuropathy, and cognitive function impairment) that reduce the efficacy of treatment. Mitochondrial dysfunction is involved in all clinical conditions including fatigue which are associated with the deficient energy metabolism of oxidative phosphorylation. Mitochondria are vulnerable to ROS which are generated endogenously (e.g. mitochondrial superoxide) and exogenously (e.g. ionizing radiation, inflammation). Once mitochondrial proteins are damaged, the affinity of substrates or enzymes is decreased resulting in mitochondrial dysfunction including reduced ATP production, increased ROS generation, and initiated apoptosis signaling. While mitochondrial dysfunction has been implicated in a variety of clinical fatigue states, the physiological pathways and pathophysiological mechanisms are complicated and remain unclear.

The primary purpose of this study is to explore the relationships between mitochondrial dysfunction and fatigue in prostate cancer patients receiving EBRT. Specific aims include: (1) identify mitochondrial-related gene expression profile changes over time; (2) quantify the severity of perceived fatigue before, during and at the end of radiation therapy; (3) determine possible pathways and early biomarkers of mitochondrial dysfunction related to fatigue in patients with prostate cancer receiving EBR. Blood samples and self-administrated questionnaires are collected at baseline, midpoint and the end of EBRT. Human mitochondrial PCR array will be utilized to identify differential regulation of genes involved in mitochondrial dysfunction at the different time points compared with gene expression from the baseline samples.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Clinically localized prostate cancer;
  2. Scheduled to receive EBRT either by 3D conformal or IMRT techniques that is not anticipated to change during the course of the study, with or without Androgen Deprivation Therapy (ADT);
  3. Able to provide written informed consent;
  4. Men greater than or equal to 18 years of age;
  5. Have enrolled in the study of molecular-genetic correlates of fatigue in cancer patients receiving localized radiation therapy (09-NR-0088).

EXCLUSION CRITERIA:

A. Any condition other than prostate cancer able to cause clinically significant fatigue including cardiovascular, pulmonary, gastrointestinal, central nervous system, psychiatric, endocrine, hematologic, renal, or immunologic disorders, and including patients with any of the following broad disease categories:

1. Systemic infections (e.g., human immunodeficiency virus [HIV], active hepatitis);
2. Documented history of major depression, bipolar disease, psychosis, or alcohol dependence/abuse within the past 5 years;
3. Uncorrected hypothyroidism and anemia;
4. Chronic inflammatory disease that may be anticipated to alter the proinflammatory cytokine profile (i.e. rheumatoid arthritis, systemic lupus erythematosus, cirrhosis).

B. Patients taking tranquilizers, steroids, and nonsteroidal anti-inflammatory agents because these medications are known to affect cytokine production;

C. Patients who have second malignancies or those receiving chemotherapy with their EBRT.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-05-24; Study Completion 2015-11-06

CONTACTS AND LOCATIONS:
Overall Officials: Leorey N Saligan, C.R.N.P., Principal Investigator — National Institute of Nursing Research (NINR)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Lemle MD. Hypothesis: chronic fatigue syndrome is caused by dysregulation of hydrogen sulfide metabolism. Med Hypotheses. 2009 Jan;72(1):108-9. doi: 10.1016/j.mehy.2008.08.003. Epub 2008 Sep 16. No abstract available. PMID 18799269
- [Background] Greenberger JS. Radioprotection. In Vivo. 2009 Mar-Apr;23(2):323-36. PMID 19414422
- [Background] Cheville AL. Cancer-related fatigue. Phys Med Rehabil Clin N Am. 2009 May;20(2):405-16. doi: 10.1016/j.pmr.2008.12.005. PMID 19389620